CLINICAL TRIAL: NCT02383641
Title: Biomarker for Wolman Disease, AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Wolman Disease (BioWolman)
Acronym: BioWolman
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BWD 06-2018
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Acid Lipase Deficiency; Acid Cholesteryl Ester Hydrolase Deficiency, Wolman Type; Cholesterol Ester Storage Disease
Keywords: Wolman disease; Biomarker
MeSH Terms: conditions — Wolman Disease; Cholesterol Ester Storage Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectometry, maximal 7,5 ml blood will be taken from the patient via using a dry blood spot filter card. To prove the correct Wolman disease diagnosis in those patients where up to the enrolment in the study no genetic testing has been done, sequencing of Wolman disease will be done. The analyses will be done at the Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Wolman disease or high-grade suspicion for Wolman disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Wolman disease blood (plasma)

DETAILED DESCRIPTION:
Wolman disease (WD) is a rare genetic disorder characterized by complete absence of an enzyme known as lysosomal acid lipase (LIPA). This enzyme is required to breakdown (metabolize) lipids in the body. Without the LIPA enzyme, lipids may abnormally accumulate in the tissues and organs of the body causing a variety of symptoms.

WD is the most severe expression of LIPA deficiency. Milder form of the disorder are known as cholesteryl ester storage deficiency. The symptoms of WD usually become apparent shortly after birth, usually during the first few weeks of life. Affected infants may develop bloating or abdominal distention and may have significant hepatosplenomegaly. Fibrosis of the liver may also occur. In some cases, fluid may accumulate in the abdominal cavity (ascites). Infants with WD have serious digestive abnormalities including malabsorption, a condition in which the intestines fail to absorb nutrients and calories from food. Malabsorption associated with WD causes persistent and often forceful vomiting, frequent diarrhea, foul-smelling, fatty stools (steatorrhea) and malnutrition. Because of these digestive complications, affected infants usually fail to grow and gain weight at the expected rate for their age and sex (failure to thrive).

Hepatosplenomegaly and protrusion of the abdomen can cause umbilical hernia, a condition in which the contents of the stomach may push through an abnormal opening or tear in the abdominal wall near the bellybutton. Additional symptoms may also occur in WD including yellowing of the skin, mucous membranes and whites of the eyes (jaundice), a persistent low-grade fever, and poor muscle tone (hypotonia). Infants may exhibit delays in the development of motor skills.

A distinct finding associated with WD is the hardening of adrenal gland tissue due to the accumulation of calcium (calcification). The adrenal glands are located on top of the kidneys and produce epinephrine and norepinephrine. Other hormones produced by the adrenal glands help to regulate the fluid and electrolyte balance in the body. Calcification of the adrenal glands is not detectable by physical examination, but can be seen with x-ray study. Calcification may prevent the adrenal glands from producing enough essential hormones and can affect metabolism, blood pressure, the immune system and other vital processes of the body.

Infants with WD may experience the loss of previously acquired skills required the coordination of muscle and motor skills (psychomotor regression). The symptoms of WD often get progressively worse eventually leading to life-threatening complications during infancy including extremely low levels of circulating red blood cells (severe anemia), hepatic dysfunction or failure, and physical wasting away and severe weakness often associated with chronic disease and marked by weight loss and loss of muscle mass (cachexia or inanition).

WD is caused by mutations of the lysosomal acid lipase (LIPA) gene. It is inherited as an autosomal recessive trait. More than 50 cases have been reported in the medical literature. However, cases may go undiagnosed or misdiagnosed making it difficult to determine the disorder's true frequency in the general population.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the plasma of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the parents before any study related procedures.
* Patients of both gender older than 2 month
* The patient has a diagnosis of Wolman disease or a high-grade suspicion for Wolman disease

High-grade suspicion present, if one or more inclusion criteria are valid:

* Positive family anamnesis for Wolman disease
* Vomiting, diarrhea
* Malnourishment, difficulty growing and gaining weight
* Enlarged liver and spleen (hepatosplenomegaly), which causes a distended abdomen
* Low muscle tone (hypotonia)
* Anemia
* x-ray reveals calcified adrenal glands

Exclusion Criteria:

* No Informed consent from the parents before any study related procedures.
* Patients of both gender younger than 2 month
* No diagnosis of Wolman disease or no valid criteria for profound suspicion of Wolman disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Wolman disease or high-grade suspicion for Wolman disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Wolman disease from blood | 24 months
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 month
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (3):
- Centogene AG, Rostock, Germany
- Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai, India
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided